CLINICAL TRIAL: NCT07085819
Title: A Prospective, Randomized, Double Blind, Placebo Controlled Study To Evaluate The Effects Of Ashwagandha (Withania Somnifera,Ws) Root Plus Leaf Aqueous Extract On Quality Of Sleep In Subjects With Non-Restorative
Brief Title: Sleep Promoting Properties of a Botanical Extract in a Population Complaining From Non-Restorative Sleep (NRS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kerry Group P.L.C (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: S24-1511769
Record Dates: First submitted 2025-07-10; First posted 2025-07-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Non Restorative Sleep; Sleep Disorder (Disorder)
Keywords: Sleep quality; Attention; Focus; Actigraph
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — PACEBO protocol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1:1:1 ratio to receive either a dose of a Botanical Extract or a placebo. Study products will be dispensed by the site according to the randomization scheme during the study visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Botanical Extract 125 (Experimental): 125 mg
  Interventions: Dietary Supplement: Botanical Extract, 125mg
- Botanical Extract 250 (Experimental): 250 mg
  Interventions: Dietary Supplement: Botanical Extract, 250mg
- Botanical Extract 500 (Experimental): 500 mg
  Interventions: Dietary Supplement: Botanical Extract, 500mg
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Pacebo

INTERVENTIONS:
Dietary Supplement: Botanical Extract, 125mg — Two capsules per day (125 mg/day) before sleep, with or without food, for 8 weeks.
  Arms: Botanical Extract 125
Dietary Supplement: Botanical Extract, 250mg — Two capsules per day (250 mg/day) before sleep, with or without food, for 8 weeks.
  Arms: Botanical Extract 250
Dietary Supplement: Botanical Extract, 500mg — Two capsules per day (500 mg/day) before sleep, with or without food, for 8 weeks
  Arms: Botanical Extract 500
Dietary Supplement: Pacebo — Two capsules per day before sleep, with or without food, for 8 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effect of the Botanical Extract in improving sleep symptoms of nonrestorative sleep (NRS) in healthy adults. The main question it aims to answer is

• Does the Botanical Extract improve sleep quality and reduce symptoms of nonrestorative sleep (NRS)? Researchers will compare the Botanical Extract to a placebo to see if it works.

Participants will:

* Take one of 3 doses of the Botanical Extract (125 mg/day, 250mg/day ,500mg/day) or a placebo every day for 8 weeks.
* Visit the clinic four times for checkups and tests and receive three follow-up phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 18 and 65 years, inclusive.
3. Self-reported unrefreshing sleep despite sufficient sleep duration for at least three nights a week over a one-month period.
4. Have a RSQ-W total score of ≤50 at screening.
5. TSH values between 0.27 - 4.20 miU/L
6. Is in general good health, as determined by the investigator.
7. Willing to consume the Study Product daily for the duration of the study.

Exclusion Criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
   2. Has a male sexual partner who is surgically sterilized prior to the Screening Visit and is the only male sexual partner for that Participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.
   5. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
3. Has a score ≥10 on Patient Health Questionnaire 8 item (PHQ-8)
4. Has a score ≥10 on Athens Insomnia Scale (AIS)
5. Participants at a high risk of sleep apnoea as determined by Berlin questionnaire/Score >5 for sleep apnoea.
6. High caffeine intake, >400mg/day
7. Has a history of drug and/or alcohol abuse at the time of enrolment.
8. Has food allergies or other issues with foods that would preclude intake of the Study Products.
9. Is an active smoker or user of nicotine products, or with a history of cigarettes smoking, tobacco or nicotine product use in the last 6 months.
10. Has undertaken shift work within the last three months or plans to undertake shift work during the study.
11. Travel across three time zones in the two months prior to screening or plans to travel across time zones during intervention.
12. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results. Excluded health conditions include:

    1. Diagnosed gastrointestinal disease.
    2. Respiratory disorders
    3. Seizure disorders
    4. Type 1 or 2 diabetes mellitus
    5. Thyroid disorders
    6. Uncontrolled hypertension
    7. Cardiovascular disease
    8. Immunocompromised health conditions
13. Current or recent (in the 12 weeks prior to screening) use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

    1. Barbiturates, anticonvulsants, benzodiazepines, neuroleptics
    2. Hypnotics
    3. Melatonin
14. Current or recent (in the 4 weeks prior to screening) use of prohibited nutritional or non-nutritional supplements, including:

    1. Herbal sleep aid supplements (St. John's Wort, Ginkgo-biloba, kava kava)
    2. Ashwagandha
    3. Caffeine supplements
15. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
16. Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sleep restorative quality | 8 weeks
  To evaluate the impact of 8 weeks daily supplementation of the Botanical Extract on Non-Restorative Sleep (NRS) as assessed by Restorative Sleep Questionnaire (RSQ-W) score compared to placebo. The total score range from 0-100 with higher scores indicating better restorative sleep.

SECONDARY OUTCOMES:
Sleep Quality | 8 weeks
  To evaluate the impact of 8 weeks daily supplementation with the Botanical Extract compared to placebo on Sleep quality as assessed by Pittsburgh Sleep Quality Questionnaire (PSQI). The total score range from 0 to 21 with the higher score indicating worse sleep quality.
Attention-Rapid Visual Information Processing (RVIP) | 8 weeks
  To evaluate the impact of 8 weeks of daily supplementation with the Botanical Extract compared to a placebo on attention using the Millisecond Rapid Visual Information Processing (RVIP) task. The following metrics will be collected and evaluated: latency (speed of response) probability of false alarms, and sensitivity
Attention-Sustained Attention to Response Task (SART). | 8 weeks
  To evaluate the impact of 8 weeks of daily supplementation with the Botanical Extract compared to a placebo on attention as assessed by the Millisecond Sustained Attention to Response Task (SART). The following metrics will be collected and evaluated: errors of commission, errors of omission, and reaction time.
Cognition | 8 weeks
  To evaluate the impact of 8 weeks daily supplementation with the Botanical Extract compared to placebo on cognition as assessed by Cognitive Function: PROMIS - Abilities-Short Form 8a. The form consists of 8 items, each rated on a 5-point scale from "Never" to "Very often" with higher scores indicating better cognitive function
Stress | 8 weeks
  To evaluate the impact of 8 weeks daily supplementation with the Botanical Extract compared to placebo on stress as assessed by serum cortisol levels (μg/dL).
Sleep parameters-Total Sleep Time (TST) | 24-hour wear time for 8 weeks
  To assess the effect of 8 weeks of daily Botanical Extract supplementation versus placebo on TST(minutes), based on Actigraphy-measured average weekly differences and total change from baseline (Day 0) to Day 56.
Sleep Parameters- Wake After Sleep Onset (WASO) | 24-hour wear time for 8 weeks
  To assess the effect of 8 weeks of daily Botanical Extract supplementation versus placebo on WASO (minutes), based on Actigraphy-measured average weekly differences and total change from baseline (Day 0) to Day 56.
Sleep Parameters- Sleep Onset Latency (SOL) | 24-hour wear time for 8 weeks.
  To assess the effect of 8 weeks of daily Botanical Extract supplementation versus placebo on SOL (minutes), based on Actigraphy-measured average weekly differences and total change from baseline (Day 0) to Day 56.
Sleep Parameters- Sleep Efficiency (SE) | 24-hour wear time for 8 weeks
  To assess the effect of 8 weeks of daily Botanical Extract supplementation versus placebo on SE (%), based on Actigraphy-measured average weekly differences and total change from baseline (Day 0) to Day 56. 24-hour wear time for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Principal Investigator — Atlantia Clinical Trials LTD.
Locations (1):
- Atlantia Food Clinical Trials Ltd., Cork, Ireland

IPD SHARING:
Plan to Share IPD: No